CLINICAL TRIAL: NCT02370901
Title: Cranial Orthotic Device Versus Repositioning Techniques for the Management of Plagiocephaly: the CRANIO Randomized Trial
Acronym: CRANIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pat Ricalde,DDS, MD, FACS (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor-Investigator, Pat Ricalde,DDS, MD, FACS, Director, Florida Craniofacial Institute, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Plagiocephaly
Record Dates: First submitted 2015-02-05; First posted 2015-02-25 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Plagiocephaly, Nonsynostotic
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic | interventions — Head Protective Devices; Home Infusion Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Helmet (Experimental): Patients will be referred to a cranial orthotist who will create a custom cranial orthotic device. They will undergo adjustments monthly. At these appointments anthropometric measurements will be done by the cranial orthotist. The orthotist will be blinded and will not be informed of which patient is involved in the study.
  Interventions: Device: Helmet
- home therapies (Experimental): Patients will be referred to a physical therapist. They will be offered education, neck stretching exercises, and repositioning techniques, and reassurance.
  Interventions: Behavioral: home therapies

INTERVENTIONS:
Device: Helmet — Custom fitting helmet, FDA approved, to allow reshaping of the infant skull
  Other Names: Cranial Orthotic Device, Starband
  Arms: Helmet
Behavioral: home therapies — parents will be instructed to do home neck stretching exercises, as well as repositioning techniques to keep baby off the flat spot. They will also be offered reassurance.
  Other Names: NSE/ RPT
  Arms: home therapies

SUMMARY:
This study evaluates the effectiveness of repositioning techniques and neck stretching exercises in comparison to cranial orthotic devices (COD) in correcting plagiocephaly in infants.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial with the goal of recruiting 226 participants. The participants will be between the ages of 4-7 months and will be randomized into two groups: Treatment group A, which will provide treatment using cranial orthotic devices (CODs) ; and Treatment group B, which will provide treatment using repositional techniques and neck stretching exercises. These participants will be offered enrollment if they have deformational molding with CVA greater than 6 mm and/or CI> 90%.

Asymmetric plagiocephaly is defined by cranial vault index (CVA). CVA is the difference between two diagonal cranial diameters (CVA= Longer diagonal-shorter diagonal). Cranial diameters are measured from orbitale superius suture to orbitale superius rear (see Appendix 1). Normal CVA is <6mm, mild CVA is 6-10mm, moderate CVA is 11-15mm, and severe CVA is >15mm. Brachycephaly is defined by the cephalic index (CI). This measurement is the width/length of cranium x100. Length of cranium is measured from glabella to opisthocranion and width is measured from eurion to eurion. Normal CI is 75-90%, mild brachycephaly is 90.1-95%, moderate brachycephaly is 95.1-100%, severe brachycephaly is >100%. Currently, repositioning exercises and helmeting therapy are both options given to the parents as there is no consensus on preferred standard of care. Once the parents have made the decision, the study investigators will monitor the patient and change therapy if there is no response to treatment or if the parents decide they would like to change therapies.

The randomization will be conducted by using a system created by the USF Department of Biostatistics. It involves a covariate adaptive randomization so that the patients will continue to be randomized throughout the trial but still allowing for covariates. Covariates for this study will be :

* type of deformity - Isolated plagiocephaly (CVA >6; 75 < CI < 90), isolated brachycephaly (CVA<6; CI > 90), and mixed brachy/ plagiocephaly (CVA > 6; CI > 90)
* severity of deformity - a CVA of 10 mm would be compared to another CVA of 10mm

Once families consent for their child to be a participant, basic demographic information will be collected. Study investigators will also collect data on developmental delay. Participants will be randomized by the physician to ensure appropriate grouping into each of the above mentioned covariates. The participants'' families will subsequently be notified the same day of the results of randomization into Treatment Group A or Treatment Group B. Both treatments are currently equally used in plagiocephaly, so there is no harm to the patient in being selected for one group versus another. The physician will re-evaluate the patients at 3 months, and if no progress is made , or if the parents are unhappy with the randomized form of treatment, the parents will have the option of switching to another group.

Potential adverse outcomes of the treatments themselves are listed as follows:

Treatment Group A (Cranial Orthotic Devices): Skin irritation due to helmeting

Treatment Group B: Pain caused by inappropriate technique in exercises

Study consent forms will include these and any other potential adverse outcomes, with a direct line to our office for notification. Benefits include correction of the plagiocephaly, and will be explained to the parents as the goal of treatment. All adverse outcomes will be reported to the IRB. Of note, these outcomes have yet to be witnessed by our staff despite years of treating patients with these methods.

Once randomized and selected, Treatment Group A will be fitted for CODs and will undergo monthly adjustments by a licensed cranial orthotist at West Coast Brace and Limb. This is standard of care for plagiocephaly. Monitoring of the patient's use of the helmet will be the responsibility of the parents, with goal of treatment to be 23 hours per day. The orthotist will have no knowledge of whether patients are enrolled in the study versus not, and will be conducting the normal responsibilities for their job. Data that is collected will be the same for all patients regardless of study enrollment. The principal study investigator, Dr. Ricalde, will be the only person with knowledge and access to the data collection for study patients during these visits.

Treatment Group B will be asked appropriate questionnaires by FCI staff and be encouraged to perform at-home repositioning techniques and neck stretching exercises. If the patient has any concerns they will be asked to come in for evaluation by a licensed physical therapist. This is the standard of care for plagiocephaly. The physical therapist will have no knowledge of whether patients are enrolled in the study versus not, and will be conducting the normal responsibilities for their job. Data that is collected will be the same for all patients regardless of study enrollment. Dr. Ricalde will be the only person with knowledge and access to the data collection for study patients during these visits.

The physical therapist and the orthotist will both be blinded to study participants, but true blinding of the treatment is not possible as the treatments require some knowledge by the parents. Initially, data will include a health questionnaire to screen for sex and developmental delay , as well as having initial CVA and CI measurements via STAR Scanner device, a standard device used by orthotists using laser light that has no harmful effects to the patient. In addition to initial measurements, patients will have measurements taken monthly (CVA and CI) by the cranial orthotist. All patients will receive photos, Star Scanner measurements, and questionnaires A and C at 6, 12, 24 months to evaluate treatment progression. Questionnaires will be administered to parents to assess satisfaction at 6, 12, 24 months. The option to switch treatment will be conducted at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with deformational molding (CVA greater than 6mm, CI > 90%, or mixed)

Exclusion Criteria:

* Children younger than 4 months and older than 7 months
* Children with plagiocephaly due to craniosynostosis, neoplasm, vertebral, or hydrocephalus.
* Scaphocephaly

Ages: 4 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-11-06 (Estimated); Study Completion 2022-11-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of helmet versus repositioning techniques for treatment of deformational molding (CVA must be less than or equal to (x-5)/2 and/or CI must be less than or equal to (x-89)/2) | 24 months
  CVA must be less than or equal to (x-5)/2 and/or CI must be less than or equal to (x-89)/2

SECONDARY OUTCOMES:
Parent satisfaction | 12 months
  questionnaire will be administered at 6, 12, 24 months
Impression of skull deformity | 24 months
  questionnaire will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Pat Ricalde, MD,DDS,FACS, Principal Investigator — Florida Craniofacial Institute
Locations (1):
- The Florida Craniofacial Institute, Tampa, Florida, United States

REFERENCES:
- [Result] van Wijk RM, Boere-Boonekamp MM, Groothuis-Oudshoorn CG, van Vlimmeren LA, IJzerman MJ. HElmet therapy Assessment in infants with Deformed Skulls (HEADS): protocol for a randomised controlled trial. Trials. 2012 Jul 9;13:108. doi: 10.1186/1745-6215-13-108. PMID 22776627